CLINICAL TRIAL: NCT05328128
Title: Investigation of the Effect of Toilet Training Given to Children Who Have no Problems in Their Social-emotional Development on the Process of Acquiring Toilet Habits
Brief Title: Investigation of the Effect of Toilet Training Given to Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hamdullah Cem Kaçmaz, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2022-03-18; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Toilet Training
Keywords: Toilet training; Social-emotional development; Child

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Children and families included in the study group were directed to the child development unit to receive toilet training.
  Interventions: Behavioral: Toilet training
- Control Group (No Intervention): The control group consisted of families who wanted to manage toilet training process themselves.

INTERVENTIONS:
Behavioral: Toilet training — As the training model, Brazelton's child-oriented toilet training method was taken as the basis in study group. In addition, literature studies on toilet training in Turkey were scanned and the final form of training to be given to mothers was created. In the control group, families manage training process themselves.
  Arms: Study Group

SUMMARY:
In the study, it was aimed to examine the factors affecting the toilet training of children aged 18-36 months who have no problems in social-emotional development and the effect of professional support on the toilet training process.

DETAILED DESCRIPTION:
Toilet training studies in Turkey and analyzes of bladder, bowel control and training completion times in these studies are limited. In this study, training processes were examined separately, and the factors that were not studied frequently until today were investigated. Also the effects of the professional support provided to children who did not have problems in social-emotional development on the process were examined.

ELIGIBILITY:
Inclusion Criteria:

* not having received toilet training
* age of the child between 18-36 months
* normal social-emotional development
* no known chronic disease

Exclusion Criteria:

* having received toilet training
* the child's age is outside the range of 18-36 months
* abnormal social-emotional development
* presence of chronic disease

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Toilet training completion age | 6 months
  It was defined as the age at which bladder and bowel control were fully achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Kara Uzun, Study Chair — University of Health Sciences, Ankara City Hospital, Children's Hospital; Sevilay Yildiz Akkus, Study Chair — University of Health Sciences, Ankara City Hospital, Children's Hospital; Bahar Cuhaci Cakir, Study Chair — Gazi University; Eda Ozaydin, Study Chair — University of Health Sciences, Ankara City Hospital, Children's Hospital
Locations (1):
- University of Health Sciences, Ankara City Hospital, Children's Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No